CLINICAL TRIAL: NCT03515304
Title: Evolocumab in Acute Coronary Syndrome: A Double-Blind Randomized Placebo Controlled Study
Brief Title: Evolocumab in Acute Coronary Syndrome
Acronym: EVACS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB00156313
Record Dates: First submitted 2018-04-10; First posted 2018-05-03 (Actual); Results first posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — evolocumab

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Persons performing the PET imaging, laboratory technicians are all masked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Evolocumab (Experimental): 420 mg evolocumab administered subcutaneously using an autoinjector/pen in NSTEMI patients within 24 hours, or one day, of admission.
  Interventions: Drug: Evolocumab
- Placebo (Placebo Comparator): Placebo administered subcutaneously using an autoinjector/pen in NSTEMI patients within 24 hours, or one day, of admission.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Evolocumab — 420 mg evolocumab administered subcutaneously using an autoinjector/pen in NSTEMI patients within 24 hours, or one day, of admission.
  Other Names: Repatha
  Arms: Evolocumab
Drug: Placebo — Placebo administered subcutaneously using an autoinjector/pen in NSTEMI patients within 24 hours, or one day, of admission.
  Arms: Placebo

SUMMARY:
Vascular and myocardial inflammation are significantly increased in Acute Coronary Syndrome (ACS) patients, are closely correlated to LDL-C levels, and are associated with these adverse consequences in the post-ACS patient population. Serum proprotein convertase subtilisin/kerin type 9 (PCSK9) levels are also increased in ACS, may raise LDL-C, and the investigators' pre-clinical studies indicate that PCSK9 is also a potent inducer of vascular inflammation. The addition of the PCSK9 antibody evolocumab, currently approved to lower LDL-C in certain patient populations, to current medical therapies would appear to be of particular benefit in an important subset of ACS patients, those with non-ST elevation myocardial infarction (NSTEMI) by markedly reducing LDL-C, stabilizing vulnerable plaque, and limiting inflammation-associated myocardial cell loss and resultant dysfunction.

DETAILED DESCRIPTION:
In a placebo-controlled, randomized double blind trial, the addition of evolocumab to standard care in NSTEMI patients (1) decreases LDL-C during hospitalization and at 30 days, (2) decreases vascular/plaque and myocardial inflammation as assessed by Positron Emission Tomography (PET) scanning at 30 days, and improves (3) serum markers of endothelial function at hospital discharge and at 30 days, and (4) echocardiographic assessment of left ventricular function at 30 days and six months.

This is the first PCSK9 inhibitor trial which examines these outcomes in the ACS patient population. It will provide valuable data on the extent and time course of LDL-C reduction as well as the impact of inhibition on inflammatory markers and on imaging assessment of vascular and myocardial inflammation, all of which may significantly impact important clinical outcomes in this high risk patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* Non ST segment elevation myocardial infarction
* Troponin I >/ 5.0 ng/dL
* Permission of attending physician

Exclusion Criteria:

* ST elevation myocardial infarction
* Patients requiring invasive hemodynamic support
* Scheduled for cardiac surgery
* Current or prior treatment with a PCSK9 antibody
* Current participation in an intervention clinical trial
* Female of childbearing potential who has not used acceptable method(s) of birth control for at least one month prior to screening
* Contraindication to statin therapy
* Subject likely not able to complete protocol related visits or procedures
* Latex allergy
* History of hypersensitivity to any monoclonal antibody

Ages: 25 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-05-20 (Actual); Primary Completion 2024-10-25 (Actual); Study Completion 2025-03-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten M Leucker, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Steven Paul Schulman, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vavuranakis MA, Jones SR, Ziogos E, Blaha MJ, Williams MS, Foran P, Schindler TH, Lai S, Schulman SP, Gerstenblith G, Leucker TM. The Trajectory of Lipoprotein(a) During the Peri- and Early Postinfarction Period and the Impact of Proprotein Convertase Subtilisin/Kexin Type 9 Inhibition. Am J Cardiol. 2022 May 15;171:1-6. doi: 10.1016/j.amjcard.2022.01.058. Epub 2022 Mar 21. PMID 35314069

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Evolocumab | Placebo
Started | 30 | 30
Completed | 30 | 27
Not Completed | 0 | 3
Not completed — Lost to Follow-up | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Placebo: placebo group
- Evolocumab: evolocumab group
- Total: Total of all reporting groups
Arm/Group | Placebo | Evolocumab | Total
Number analyzed (Participants) | 30 | 30 | 60
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 19 | 18 | 37
  >=65 years | 11 | 12 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (13.9) | 59.4 (14.2) | 60.1 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 9 | 25
  Male | 14 | 21 | 35
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 11 | 8 | 19
  White | 16 | 20 | 36
  More than one race | 3 | 1 | 4
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 30 | 30 | 60

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in LDL-Cholesterol
Time Frame: Baseline to 30 days
Population: Participants with data collected
Measure: Median (Inter-Quartile Range); unit: percent change
Arm/Group | Evolocumab | Placebo
Number analyzed (Participants) | 30 | 27
percent change | -68.78 [-76.24 to -46.82] | -27.58 [-46.46 to 1.38]

2. Primary Outcome: Change From Baseline in Target to Background Ratio Fluorodeoxyglucose (FDG) Positron Emission Tomography (PET) Scans
Description: PET Imaging for Inflammation: Change from baseline in target to background ratio Fluorodeoxyglucose (FDG) PET scans in the myocardium.
Time Frame: Baseline to 30 days
Population: Participants with PET data collected and adequate image quality for analysis
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Evolocumab | Placebo
Number analyzed (Participants) | 25 | 30
ratio | -26.7 (20.4) | -10.4 (36.2)

3. Secondary Outcome: Change in Left Ventricular Volume as Assessed by Echocardiography
Description: Evaluation of left ventricular volume (ml) by echocardiography
Time Frame: Baseline, day 30 and 6 months
Reporting Status: Not Posted

4. Secondary Outcome: Change in Ejection Fraction as Assessed by Echocardiography
Description: Evaluation of ejection fraction (%) by echocardiography
Time Frame: Baseline, day 30 and 6 months
Reporting Status: Not Posted

5. Secondary Outcome: Change in Plasma Proprotein Convertase Subtilisin Kexin-9 (PCSK9) Levels (ng/ml)
Description: Change from baseline in PCSK9 serum levels
Time Frame: Baseline, day 30 and 6 months
Reporting Status: Not Posted

6. Secondary Outcome: Change in Plasma Soluble Lectin-like Oxidized Low-density Lipoprotein Receptor-1 (LOX-1)
Description: Change from baseline in plasma soluble lectin-like oxidized low-density lipoprotein receptor-1 (LOX-1) (pg/ml)
Time Frame: Baseline, day 30 and 6 months
Reporting Status: Not Posted

7. Secondary Outcome: PET-FDG Assessed Vascular Inflammation as Assessed by Standardized Uptake Value (SUV)
Description: Target artery to background ratio endpoint (standardized uptake value) for left carotid artery
Time Frame: Baseline to day 30
Population: Participants with PET data collected and adequate image quality for analysis
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | Evolocumab | Placebo
Number analyzed (Participants) | 20 | 14
SUV | 3.134705882 (8.448074995) | 3.708333333 (10.05850912)
Statistical Analysis 1: Comparison: Evolocumab vs Placebo; Test type: Superiority; p = 0.2497, t-test, 2 sided

8. Secondary Outcome: Change in New York Heart Association (NYHA) Class
Description: Assess NYHA class I-IV
Time Frame: Baseline, day 30 and 6 months
Reporting Status: Not Posted

9. Secondary Outcome: Change in High Sensitivity C-reactive Protein (Hs-CRP) Serum Levels
Description: Change from baseline in hs-CRP serum levels (mg/L)
Time Frame: Baseline, day 30 and 6 months
Reporting Status: Not Posted

10. Secondary Outcome: Change in Tumor Necrosis Factor (TNF)-Alpha Serum Levels
Description: Change from baseline in TNF-alpha serum levels (pg/mL)
Time Frame: Baseline, day 30 and 6 months
Reporting Status: Not Posted

11. Secondary Outcome: Change in Plasma Levels of Interleukin 1
Description: Change from baseline in serum levels of Interleukin 1 (pg/mL)
Time Frame: Baseline, day 30 and 6 months
Reporting Status: Not Posted

12. Secondary Outcome: Change in Serum Levels of Interleukin 6
Description: Change in baseline in serum levels of Interleukin 6 (pg/mL)
Time Frame: Baseline, day 30 and 6 months
Reporting Status: Not Posted

13. Secondary Outcome: Change in Serum Levels of Interleukin 10
Description: Change in baseline in serum levels of Interleukin 10 (pg/mL)
Time Frame: Baseline, day 30 and 6 months
Reporting Status: Not Posted

14. Secondary Outcome: Change in Canadian Angina Class
Description: Assess Canadian Angina Classification, I-IV
Time Frame: Baseline, 30 days, 6 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: from enrollment through 30-day follow-up
Arm/Group | Evolocumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 2/30 | 6/30
Other Adverse Events (participants affected / at risk) | 13/30 | 6/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evolocumab (N=30) | Placebo (N=30)
Acute kidney injury requiring intermittent hemodialysis (Renal and urinary disorders) | 0 (0) | 1 (1)
Gastrointestinal bleed (Gastrointestinal disorders) | 0 (0) | 1 (1)
Recurrent non-ST elevation myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Transient myocardial ischemia prompting hospitalization (Cardiac disorders) | 1 (1) | 0 (0)
Hospitalization for planned vascular surgery (Vascular disorders) | 1 (1) | 0 (0)
Hospitalization for neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Transient ischemic attack, slurred speech (Nervous system disorders) | 0 (0) | 1 (1)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Evolocumab (N=30) | Placebo (N=30)
Angina (Cardiac disorders) | 2 (2) | 2 (2)
Pre-syncope (Nervous system disorders) | 1 (1) | 0 (0)
Ecchymosis injection site (Skin and subcutaneous tissue disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1)
Post-infarction pericarditis (Cardiac disorders) | 1 (1) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-06-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT03515304/Prot_SAP_000.pdf